CLINICAL TRIAL: NCT01201551
Title: Effect of Alphagan and Xalatan Eye Drops on Corneal Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 088-Mom-2010
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Primary Vascular Dysregulation
Keywords: Alphagan; Xalatan; corneal temperature; primary vascular dysregulation
MeSH Terms: interventions — Brimonidine Tartrate; Latanoprost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy subjects without PVD (Active Comparator): healthy subjects without primary vascular dysregulation Intervention: Brimonidine, Latanoprost and Placebo
  Interventions: Drug: Brimonidine; Drug: Latanoprost; Drug: Placebo
- healthy subjects with PVD (Active Comparator): healthy subjects with primary vascular dysregulation Intervention: Brimonidine, Latanoprost and Placebo
  Interventions: Drug: Brimonidine; Drug: Latanoprost; Drug: Placebo

INTERVENTIONS:
Drug: Brimonidine — Week1, day2: 1 eyedrop/right eye Week2, day1: 1 eyedrop/left eye Week2, day2: 1 eyedrop/left eye
  Other Names: Alphagan
Drug: Latanoprost — Week1, day1: 1 eyedrop/right eye Week1, day2: 1 eyedrop/right eye Week2, day2: 1 eyedrop/left eye
  Other Names: Xalatan
Drug: Placebo — Week1, day1: 1 eyedrop/left eye Week1, day2: 2 eyedrops/left eye Week2, day1: 1 eyedrop/right eye Week2, day2: 2 eyedrops/right eye
  Other Names: Fermavisc

SUMMARY:
It is already known that the local treatment with Alphagan eye drops (a drug commonly used by glaucoma patients) reduces ocular blood flow. In-vitro studies suggest that the vasoconstrictive effect of Alphagan is more pronounced when this drug is combined with a prostaglandin analogue (eg. Xalatan eye drops). The investigators also question whether this effect is more pronounced in subjects suffering from a primary vascular dysregulation (PVD). To test for the effect of these drugs on PVD and non-PVD subjects the investigators will take measurements of corneal temperature as surrogate for ocular blood flow.

DETAILED DESCRIPTION:
The investigators would like to investigate the effect of Alphagan eye drops, Xalatan eye drops and their combination (both Alphagan and Xalatan) on corneal temperature in healthy subjects with and without a primary vascular dysregulation (PVD).

The investigators would like to answer the following questions:

1. Do the individual drugs influence the circulation to the eye as quantified indirectly via corneal temperature?
2. Does the combination of Alphagan and Xalatan give an additive or even potentiated effect?
3. Is the sequence of application of drugs of relevance (Alphagan applied first, Xalatan second, or vice versa)?
4. Do PVD and non-PVD subjects respond differently to these drugs?

20 healthy non-PVD subjects and 20 healthy PVD subjects in the age range from 20-40 years will be recruited. Recruited subjects will have all measurements: corneal temperature, intraocular pressure (IOP), ear temperature, blood-pressure. Both prior to and after instillation of eye drops (Xalatan, Alphagan and placebo).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 18-48 years
* normal findings on ophthalmological examination

Exclusion Criteria:

* history of ocular or systemic disease
* chronic or current systemic or topical medication
* drug or alcohol abuse
* art. hypertension

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Corneal temperature | Week 1: day 1 and 2 before eyedrops and after. Week 2: day 1 and 2 before eyedrops and after.

SECONDARY OUTCOMES:
Intraocular pressure | Week 1: day 1 and 2 before eyedrops and after. Week 2: day 1 and 2 before eyedrops and after.
Ear temperature | Week 1: day 1 and 2 before eyedrops and after. Week 2: day 1 and 2 before eyedrops and after.
Blood pressure | Week 1: day 1 and 2 before eyedrops and after. Week 2: day 1 and 2 before eyedrops and after.

CONTACTS AND LOCATIONS:
Overall Officials: Josef Flammer, MD, Study Director — University of Basel, Dept. of Ophthalmology
Locations (1):
- University of Basel, Dept. of Ophthalmology, Basel, Switzerland